CLINICAL TRIAL: NCT02684734
Title: Prevalence of Cytomegalovirus Infection in Patients With Quiescent Ulcerative Colitis
Acronym: PROVE-UC
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brian Bressler, Clinical Associate Professor of Medicine, University of British Columbia
Other Study IDs: H15-00197
Record Dates: First submitted 2016-01-27; First posted 2016-02-18 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis; Cytomegalovirus Infections
Keywords: Ulcerative Colitis; UC; Cytomegalovirus; CMV
MeSH Terms: conditions — Colitis, Ulcerative; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients on no immunosuppressant: This includes patients on no medication or mesalamine.
- Patients on immunosuppressants: This includes patients on biologics, azathioprine (AZA), 6-mercaptopurine (6-MP), or corticosteroid. These patients will be sub-analyzed to: a) Patients on one immunosuppressive therapy with AZA, 6-MP, biologic or corticosteroid; b) Patients on combination therapy with AZA or 6-MP and biologic; c) Patients on triple therapy with corticosteroid, AZA or 6-MP, and biologic; d) Patients on corticosteroid and one other immunosuppressive therapy such as AZA, 6-MP, or biologic.

SUMMARY:
Colitis from reactivation of established cytomegalovirus (CMV) colonization can complicate the clinical course in patients with an acute flare of ulcerative colitis (UC). Accurate and timely detection of active CMV infection or disease with appropriate anti-viral therapy may reduce complications associated with acute UC flare. Limited information is available on the presence of colonic CMV infection in patients with quiescent ulcerative colitis. Prospective studies on factors associated with reactivation of CMV infection during active UC flare and its impact on disease progression are lacking.

The hypothesis of this study are as follows: 1) CMV infection is prevalent in patients with ulcerative colitis irrespective of disease severity; 2) The degree of immunosuppression directly impacts CMV infection status in patients with ulcerative colitis

DETAILED DESCRIPTION:
This is cross sectional study at St. Paul's Hospital, a tertiary academic teaching hospital. Subjects ages 19 or greater with quiescent ulcerative colitis present for routine elective surveillance endoscopy will be invited for the study.

At enrollment, subjects will be evaluated for clinical and endoscopic disease severity using Mayo score. To be eligible for the study, Mayo score must be <2. Supplemental blood tests, diagnostic test to determine CMV status, physical examination for extra-intestinal manifestation of CMV and inflammatory bowel disease, and surveillance colonoscopy with colonic biopsy will be done.

Patients will be followed longitudinally. Patients will be contacted every three months via their preferred method (telephone or email) until disease flare (clinical partial Mayo Score > 2) or one year from enrolment. Patients will be asked to contact study coordinator when they are experiencing UC flare.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 19 or greater with quiescent ulcerative colitis present for routine elective surveillance endoscopy
* At enrolment: clinical partial Mayo score < 2 prior to endoscopic evaluation
* At endoscopy: endoscopic Mayo score < 2

Exclusion Criteria:

* Patient age less than 19
* Clinical partial Mayo score at enrollment ≥ 2
* Endoscopic Mayo score ≥ 2
* Overall Mayo score > 5
* Patients with known current or previous CMV infection
* Patients with HIV, solid organ or bone marrow transplantation, immunoglobulin deficiency, and who are otherwise immunosuppressed for reasons other than treatment of ulcerative colitis, or
* Pregnant patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ulcerative colitis presenting for routine elective surveillance endoscopy will be approached for enrolment. Patients will be evaluated by the gastroenterologist at pre-endoscopy clinic visit for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of CMV infection (ie previous CMV exposure or existing CMV virus) in patients with quiescent UC undergoing routine surveillance endoscopy | upon enrollment

SECONDARY OUTCOMES:
Prevalence of cytomegalovirus (CMV) viremia (ie. active virus in bloodstream) in patients with quiescent UC receiving immunosuppressive therapy | upon enrollment
  This will be measured by serum immunoglobulin M (IgM)
Prevalence of CMV (ie. inactive virus in bloodstream) in patients with quiescent UC receiving immunosuppressive therapy | 1 year
  This will be measured by serum immunoglobulin G (IgG)
Prevalence of CMV viremia in patients with quiescent UC receiving immunosuppressive therapy | 1 year
  This will be measured by viral load in the serum.
Prevalence of cytomegalovirus (CMV) infection of the colon in patients with quiescent UC receiving immunosuppressive therapy. | 1 year
  This will be measured by colonic biopsy CMV polymerase chain reaction (PCR)
Prevalence of CMV infection of the colon in patients with quiescent UC receiving immunosuppressive therapy. | 1 year
  This will be measured histopathologically with CMV immunochemistry staining.
Correlation of serum CMV status with colonic CMV manifestation in patients with quiescent UC | upon enrollment
Correlation of serum CMV status with colonic CMV manifestation in patients with known latent CMV infection during active UC flare | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, Principal Investigator — Division of Gastroenterology, Department of Medicine St. Paul's Hospital, Vancouver, BC, Canada
Locations (1):
- GI Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayre K, Warren BF, Jeffery K, Travis SP. The role of CMV in steroid-resistant ulcerative colitis: A systematic review. J Crohns Colitis. 2009 Sep;3(3):141-8. doi: 10.1016/j.crohns.2009.03.002. Epub 2009 Apr 14. PMID 21172262
- [Background] Domenech E, Vega R, Ojanguren I, Hernandez A, Garcia-Planella E, Bernal I, Rosinach M, Boix J, Cabre E, Gassull MA. Cytomegalovirus infection in ulcerative colitis: a prospective, comparative study on prevalence and diagnostic strategy. Inflamm Bowel Dis. 2008 Oct;14(10):1373-9. doi: 10.1002/ibd.20498. PMID 18452205
- [Background] Dimitroulia E, Spanakis N, Konstantinidou AE, Legakis NJ, Tsakris A. Frequent detection of cytomegalovirus in the intestine of patients with inflammatory bowel disease. Inflamm Bowel Dis. 2006 Sep;12(9):879-84. doi: 10.1097/01.mib.0000231576.11678.57. PMID 16954807
- [Background] Kim YS, Kim YH, Kim JS, Cheon JH, Ye BD, Jung SA, Park YS, Choi CH, Jang BI, Han DS, Yang SK, Kim WH; IBD Study Group of the Korean Association for the Study of Intestinal Diseases. The prevalence and efficacy of ganciclovir on steroid-refractory ulcerative colitis with cytomegalovirus infection: a prospective multicenter study. J Clin Gastroenterol. 2012 Jan;46(1):51-6. doi: 10.1097/MCG.0b013e3182160c9c. PMID 21552140
- [Background] Kishore J, Ghoshal U, Ghoshal UC, Krishnani N, Kumar S, Singh M, Ayyagari A. Infection with cytomegalovirus in patients with inflammatory bowel disease: prevalence, clinical significance and outcome. J Med Microbiol. 2004 Nov;53(Pt 11):1155-1160. doi: 10.1099/jmm.0.45629-0. PMID 15496396
- [Background] Roblin X, Pillet S, Oussalah A, Berthelot P, Del Tedesco E, Phelip JM, Chambonniere ML, Garraud O, Peyrin-Biroulet L, Pozzetto B. Cytomegalovirus load in inflamed intestinal tissue is predictive of resistance to immunosuppressive therapy in ulcerative colitis. Am J Gastroenterol. 2011 Nov;106(11):2001-8. doi: 10.1038/ajg.2011.202. Epub 2011 Jul 26. PMID 21788989
- [Background] Sipponen T, Turunen U, Lautenschlager I, Nieminen U, Arola J, Halme L. Human herpesvirus 6 and cytomegalovirus in ileocolonic mucosa in inflammatory bowel disease. Scand J Gastroenterol. 2011 Nov;46(11):1324-33. doi: 10.3109/00365521.2011.605466. Epub 2011 Aug 31. PMID 21879802
- [Background] Yoshino T, Nakase H, Ueno S, Uza N, Inoue S, Mikami S, Matsuura M, Ohmori K, Sakurai T, Nagayama S, Hasegawa S, Sakai Y, Chiba T. Usefulness of quantitative real-time PCR assay for early detection of cytomegalovirus infection in patients with ulcerative colitis refractory to immunosuppressive therapies. Inflamm Bowel Dis. 2007 Dec;13(12):1516-21. doi: 10.1002/ibd.20253. PMID 17828781
- [Background] McCurdy JD, Enders FT, Jones A, Killian JM, Loftus EV Jr, Bruining DH, Smyrk TC. Detection of Cytomegalovirus in Patients with Inflammatory Bowel Disease: Where to Biopsy and How Many Biopsies? Inflamm Bowel Dis. 2015 Dec;21(12):2833-8. doi: 10.1097/MIB.0000000000000556. PMID 26273816